CLINICAL TRIAL: NCT02428829
Title: Does Rapid Mobilisation as Part of an Enhanced Recovery Pathway Improve Length of Stay, Return to Function and Patient Satisfaction Post Primary Total Hip Arthroplasty?
Brief Title: Does Rapid Mobilisation Improve Length of Stay and Outcomes Post THR
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPID-1
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Arthroplasty, Replacement, Hip; Hip Replacement, Total
Keywords: hip; replacement; arthroplasty; total; orthopaedic; rehabiliation; physiotherapy; therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group will be seen by a physiotherapist to attempt walking from 4 hours post operatively, on the day of their surgery.
  Interventions: Procedure: Attempt walking from 4 hours post operatively, on the day of their surgery.
- Control (Active Comparator): Control group will receive standard physiotherapy in line with current hospital protocol including first walking approximately 24 hours post operatively
  Interventions: Procedure: Control - standard treatment

INTERVENTIONS:
Procedure: Attempt walking from 4 hours post operatively, on the day of their surgery. — Intervention group will be seen by a physiotherapist to attempt walking from 4 hours post operatively, on the day of their surgery.
  Arms: Intervention
Procedure: Control - standard treatment — standard physiotherapy in line with current hospital protocol including first walking approximately 24 hours post operatively.
  Arms: Control

SUMMARY:
This study looks to examine the effect of attempting initial postoperative walking with a patient following a total hip replacement. Currently patients rest in bed for approximately 24 hours following their operation before walking. The intervention group would aim to commence walking at between 4-6 hours after their operation.

Outcome measures to be examined would be: length of hospital stay, patient experience of physiotherapy treatment, the time taken for patients to reach functional milestones and number of postoperative medical complications.

The study is designed as a randomised controlled trial where participants would be separated randomly into two groups. One group would form the intervention group and start physiotherapy and attempted walking 4-6 hours after their operation. The other group would form the control group and would remain on the current standard rehabilitation protocol.

DETAILED DESCRIPTION:
As part of this study, patients who are waiting for a total hip replacement, and have no other serious medical problems will be given an information sheet about the study at the preoperative education group session approximately 12 weeks prior to their surgery. If they are interested they would be asked on the day of their operation if they would like to take part in the study, potential participants will have had the opportunity to ask any questions to a senior member of the research team over the telephone or at a further study specific appointment if they wish before this stage.

Any patients who agree to take part would be free to withdraw from the study at any time, without any implications for their ongoing medical treatment. Patients do not have to give a reason as to why they would like to stop taking part, this is explained during the consent process but will be reiterated to participants during the study.

Once participants have entered the study, they would be selected at random to one of two groups:

Group 1: (Rapid Mobilisation Group) Participants will be seen between 4 and 6 hours after returning to the ward after surgery. The physiotherapist would aim to start walking with them at this stage, as long as the physiotherapist feels that this is safe.

Group 2: (Control Group) Participants will be seen between 4 and 6 hours after returning to the ward after surgery. The physiotherapist would start exercises on the bed with these patients. This is standard practice and is the current patient protocol at the Royal Bournemouth Hospital. The rest of their stay as a patient would continue as normal in accordance with standard care.

The following items will be measured for each patient:

1. How long they stay in hospital after their operation
2. How satisfied they were with physiotherapy.
3. Their pain levels when walking for the first time.
4. How quickly they return to independence with walking and other tasks.
5. Whether they had any medical complications after their operation.

The null hypothesis is that rapid walking following total hip replacement does not affect the amount of time patients stay in hospital, the amount of time taken to reach functional milestones such as walking or stairs, and how the patient grades their experience of physiotherapy.

The results of this research would then be analysed both at half way through data collection and at the end of data collection by the research team and the Sponsor and would be published as part of a research paper in a medical journal. This type of study design has been chosen to provide the research team with a high quality comparison between the two groups. Due to the nature of the treatment it was felt that it wasn't possible to implement any participant or clinician blinding to the methodology.

However, both groups of patients will be treated using a treatment protocol to limit any differences between group interventions.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed written consent
* Able to understand verbal and written communication in English
* Over 18 years of age
* Primary Uni-lateral Total Hip Replacement (THR)
* No intra-operative complications
* Weight bearing status:
* Fully Weight Bearing
* Weight Bearing as Tolerated.
* Adequate home support to facilitate timely discharge.

Exclusion Criteria:

* No current or historical serious co-morbidities:
* Cerebro-Vascular Accident (CVA)
* Myocardial Infarction (MI)
* Pulmonary Embolism (PE)
* Deep Vein Thrombosis (DVT) o Diabetes Mellitus (DM)
* Significant intra or post-operative wound ooze
* Poor pre-morbid mobility/level of function (House or wheelchair bound)
* Clinical signs of DVT or PE
* Altered Weight-Bearing status
* Repair to abductor muscle complex
* Nerve block as part of anaesthetic
* Participation in any other research trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Length of inpatient hospital stay following return to the ward after total hip replacement | 7 days
  This is measured in number of days. The study would determine a change in length of stay by one day clinically significant.

SECONDARY OUTCOMES:
Patient satisfaction with physiotherapy care following completion of physiotherapy care as measured by completion of patient satisfaction questionnaire results | 12 weeks
  No significant differences between the groups or better would be considered clinically significant
Time taken for patients to reach functional milestones postoperatively | 4 hours
  An average reduction of greater than or equal to 4 hours would be considered clinically significant
The incidence rate of postoperative complications | 12 weeks
  No significant differences between the groups or better would be considered clinically significant
Numerical pain scores for the patients postoperative pain | 12 weeks
  No significant differences between the groups or better would be considered clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Efford, BSc(Hons), Principal Investigator — Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust
Locations (1):
- The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, Dorset, United Kingdom